CLINICAL TRIAL: NCT03336450
Title: A Phase 3, Multicenter, Open-label Extension Study of Buccally Administered MHOS/SHP615 in Pediatric Patients With Status Epilepticus (Convulsive) in Community Settings
Brief Title: Study of Midazolam Hydrochloride Oromucosal Solution (MHOS/SHP615) in Pediatric Patients With Status Epilepticus (Convulsive) in the Community Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP615-302
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-08

CONDITIONS: Nervous System Diseases
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHP615 (Experimental): Participants will receive a single age-specific dose (approximately 0.25 to 0.5 milligram per kilogram [mg/kg] as midazolam) of SHP615 oromucosal solution through buccal route upon onset of seizures.
  Interventions: Drug: SHP615; Drug: MHOS/SHP615

INTERVENTIONS:
Drug: SHP615 — SHP615 oromucosal solution will be administered as a single age-specific dose (2.5, 5, 7.5 and 10 mg).
  Other Names: MHOS; Midazolam hydrochloride oromucosal solution
Drug: MHOS/SHP615 — MHOS/SHP615

SUMMARY:
The purpose of this study is to determine if the investigational treatment, MHOS/SHP615, is safe and effective in children with status epilepticus (SE) (convulsive) in the community setting. This study is open-label extension for patients who completed the SHP615-301 study and who tolerated and responded to MHOS/SHP615 treatment in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the SHP615-301 study and who tolerated and responded to treatment with MHOS/SHP615 in the hospital and/or emergency room, and are considered stable for discharge from the hospital.
* Subjects who are greater than (>) 6 months and less than (<) 18 years of age at the time of investigational product administration. If the subject's exact age is not known, the subject should be excluded.
* Parent, guardian, or legally authorized representative of the child who provides informed consent and assent (when applicable) to participate in the study after initial stabilization of the subject with SE in hospital or emergency room during the SHP615-301 study. The subject also provides informed consent prior to participation, where applicable.
* Parent, guardian, or legally authorized representative who have received appropriate training/education and are deemed qualified by the investigator and are willing to:

  1. Properly administer MHOS/SHP615.
  2. Record seizure information and dosing of MHOS/SHP615 in a subject diary (including time of seizure onset, type of seizure, time necessary to administer MHOS/SHP615, time between MHOS/SHP615 administration to seizure cessation, etc.)
  3. Follow the necessary instructions to secure the safety of the subject.
* Subjects who experience generalized tonic-clonic SE with seizures accompanied by loss of consciousness with any of the following characteristics persistent at the time of study drug administration:

  1. Currently presenting with seizure (convulsive) activity and 3 or more convulsions within the preceding hour
  2. Currently presenting with seizure (convulsive) and 2 or more convulsions in succession without recovery of consciousness.
  3. Currently presenting with a single seizure (convulsive) persisting greater than or equal to (>=) 5 minutes.

Exclusion Criteria:

* Female subjects who are pregnant, suspected to be pregnant, or nursing.
* Subjects with major trauma, not necessarily restricted to the head, as the cause of the seizure.
* Subjects with known or suspected recurrent seizures due to illegal drug or alcohol withdrawal.
* Subjects with seizures due to illegal drug or acute alcoholic intoxication.
* Subjects with seizures of psychogenic origin.
* Subjects with seizures due to severe encephalitis or meningitis, as determined by the PI
* Subjects with known history of hypersensitivities, nonresponsiveness or contraindications to benzodiazepines (that is (ie), clinically significant respiratory depression, severe acute hepatic failure, myasthenia gravis, syndrome of sleep apnea, glaucoma with closed angle, or use of concomitant drugs determined by the investigator to have a contraindication to the use of benzodiazepines.)
* Subjects with a known history of benzodiazepine abuse.
* Subjects who have not responded to previous administrations of midazolam systemic therapies, including MIDAFRESA and/or DORMICUM.
* Subjects who need emergent surgical intervention and general anesthesia/intubation.
* Subjects who have been receiving human immunodeficiency virus (HIV) protease inhibitors or HIV reverse transcriptase inhibitors.
* Subjects with severe cerebral anoxia (except cerebral palsy), in the judgment of the healthcare provider.
* Have used an investigational product or been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
* Subject has prior placement of a vagus nerve stimulator.

Ages: 6 Months to 216 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas
Locations (23):
- Japan (23):
  - Yamanashi Prefectural Central Hospital, Kofu, Fujimi
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - NHO Minami-Okayama Medical Center, Okayama, Okayama-ken
  - Tokyo Women's Medical University Yachiyo Medical Center, Yachiyo, Owada Shinden
  - Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Fukuoka Children's Hospital(NW), Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - NHO Hokkaido Medical Center, Hokkaidō
  - Kumamoto Saishunso National Hospital, Kumamoto
  - NHO Nagasaki Medical Center, Nagasaki
  - NHO Nishi Niigata Chuo National Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Nakano Children's Hospital, Osaka
  - Osaka Women's and Children's Hospital(NW), Osaka
  - Aichi Children's Health and Medical Center(NW), Ōbu
  - Saitama Children's Medical Center(NW), Saitama
  - Jichi Children's Medical Center Tochigi, Saitama-shi
  - Osaka University Hospital, Suita
  - Tokyo Women's Medical University Hospital, Tokyo
  - National Center Hospital, NCNP, Tokyo
  - Tottori University Hospital, Tottori
  - Osaka University Hospital, Yamadaoka
  - Kanagawa Children's Medical Center(NW), Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Shire provides access to the de-identified individual participant data for eligible studies to aid qualified researchers in addressing legitimate scientific objectives. These IPDs will be provided following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.shiretrials.com website. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://www.shiretrials.com/en/our-commitment-to-transparency/data-sharing-with-researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in Japan between 23 April 2018 (first participant first visit) and 13 October 2020 (last participant last visit).
Pre-assignment Details: A total of 12 participants were screened, of which 9 participants were screen failures and withdrawn prior to randomization. Only 3 participants were enrolled to receive treatment and completed the study.
Groups:
- SHP615: Participants received single fixed age-specific dose (6 months to less than [<] 1 year received 2.5 milligrams [mg]; 1 to < 5 years received 5 mg; 5 to <10 years received 7.5 mg and 10 to < 18 years received 10 mg) of midazolam hydrochloride oromucosal solution (MHOS)/SHP615 buccally by caregivers on Day 1.
Period: Overall Study
Arm/Group | SHP615
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who had received a single dose of Investigational product (IP), regardless of whether the study drug administration was documented to be complete or not on the study drug administration electronic case report form (eCRF).
Arm/Group | SHP615
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.07 (1.570)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Number of Participants With Therapeutic Success
Description: Therapeutic success was defined as cessation of visible seizure activity within 10 minutes and sustained absence of visible seizure activity for 30 minutes following a single dose of SHP615 without the need for additional rescue medication. Number of participants with therapeutic success were reported.
Time Frame: From start of study drug administration up to 30 minutes post-dose
Population: Full analysis set (FAS) consisted of all participants in the safety set who had at least 1 assessment for determination of therapeutic success (cessation of seizure within 10 minutes with sustained absence of seizure for 30 minutes) performed after the administration of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Efficacy: Number of Participants Who Had Sustained Absence of Seizure Activity for at Least 1, 4, and 6 Hours
Description: Number of participants whose seizure event stopped within 10 minutes of single dose administration of SHP615 and who had sustained absence of seizure activity for at least 1, 4, and 6 hours were reported.
Time Frame: From start of study drug administration up to 1, 4, and 6 hours post-dose
Population: FAS consisted of all participants in the safety set who had at least 1 assessment for determination of therapeutic success (cessation of seizure within 10 minutes with sustained absence of seizure for 30 minutes) performed after the administration of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants
  Sustained absence for at least 1 hour | 3
  Sustained absence for at least 4 hour | 0
  Sustained absence for at least 6 hour | 1

3. Secondary Outcome: Efficacy: Time to Resolution of Seizures (Convulsions)
Description: Time to resolution of seizures (convulsions) was calculated as time from SHP615 administration to the end of the initial seizure or administration of rescue anticonvulsant medication, whichever occurs first. The initial seizure refers to the seizure which triggered the use of the IP. Participant wise data was reported for this outcome.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: FAS consisted of all participants in the safety set who had at least 1 assessment for determination of therapeutic success (cessation of seizure within 10 minutes with sustained absence of seizure for 30 minutes) performed after the administration of IP. Here, number analyzed signifies participants who were evaluable for this specific category.
Measure: Number; unit: Minutes
Arm/Group | SHP615
Number analyzed (Participants) | 3
Minutes
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 5

4. Secondary Outcome: Efficacy: Time to Recovery of Consciousness
Description: Time to recovery of consciousness in minutes was calculated only for participants who lost consciousness pre-dose as time from SHP615 administration to recovery of consciousness post-dose or administration of rescue anticonvulsant medication, whichever occurs first. Participant wise data was reported for this outcome.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 3
Measure: Number; unit: Minutes
Arm/Group | SHP615
Number analyzed (Participants) | 3
Minutes
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 4
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 143
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 5

5. Secondary Outcome: Efficacy: Percentage of Participants Who Required Additional Anticonvulsant Medication for Ongoing Status Epilepticus (SE) 10 Minutes After Administration of SHP615
Description: Percentage of participants who required additional anticonvulsant medication for ongoing SE according to the participating hospital protocol or guideline, 10 minutes after the administration of SHP615 were reported.
Time Frame: 10 minutes post-dose
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Percentage of participants | 0

6. Secondary Outcome: Efficacy: Percentage of Participants Who Failed to Respond to Treatment With SHP615
Description: Treatment failure/non-responder was defined as continuing seizure activity and/or the need for any additional rescue medication according to the participating healthcare setting protocol or guideline 10 minutes after administration of SHP615 was reported.
Time Frame: 10 minutes post-dose
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Percentage of participants | 0

7. Primary Outcome: Safety: Number of Participants With Respiratory Depression
Description: Respiratory depression, included the following measures within 24 hours after administration of the IP: i) Persistent decrease in oxygen saturation to <92 percent (%) measured up to 24 hours post-dose (i.e., <92% on room air for 2 minutes or more after dosing while monitoring [per healthcare setting protocol and/or the clinical judgment of the physician]. ii) Increase in respiratory effort such that assisted ventilation is used (bag-valve-mask ventilation or endotracheal intubation). Number of participants with respiratory depression were reported.
Time Frame: Up to 24 hours post-dose
Population: Safety set consisted of all participants who had received a single dose of IP, regardless of whether the study drug administration was documented to be complete or not on the study drug administration eCRF.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

8. Secondary Outcome: Safety: Number of Participants With Aspiration Pneumonia Reported as Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs was defined as adverse events (AEs) whose onset occurs, severity worsens or intensity increases on or after the date of SHP615 administration. Number of participants with aspiration pneumonia identified as TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Safety: Number of Participants Analyzed for Sedation or Agitation Measured by the Riker Sedation-Agitation Scale
Description: Sedation-Agitation was assessed, using the "Riker Sedation-Agitation Scale" (SAS) by the following 7-point scale: 7. dangerous agitation; 6. very agitated; 5. agitated; 4. calm, cooperative; 3. sedated; 2. very sedated; 1. unarousable. Number of participants analyzed for sedation or agitation measured by the riker sedation-agitation scale were reported.
Time Frame: 1, 4, 6, and 24 hours post-dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants
  Participant with unarousable | 0
  Participant with very sedated | 1
  Participant with sedated | 1
  Participant with calm and cooperative | 3
  Participant with agitated | 1
  Participant with very agitated | 0
  Participant with dangerous agitation | 0

10. Secondary Outcome: Safety: Number of Participants With Buccal Irritation Reported as Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs was defined as AEs whose onset occurs, severity worsens or intensity increases on or after the date of IP administration. Buccal cavity was examined for redness, inflammation and ulceration. Number of participants with buccal irritation reported as TEAEs were reported.
Time Frame: Up to 6 hours post-dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

11. Secondary Outcome: Safety: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs was defined as AEs whose onset occurs, severity worsens or intensity increases on or after the date of IP administration. Number of participants with TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Day 8)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 2

12. Secondary Outcome: Safety: Number of Participants With Clinically Significant Change in Vital Signs Reported as TEAEs
Description: Vital sign assessments included blood pressure, pulse, respiratory rate and body temperature. Any change in vital signs which were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: From start of study drug administration up to 24 hours post-dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

13. Secondary Outcome: Safety: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters Reported as TEAEs
Description: Clinical laboratory evaluations included biochemistry, endocrinology, hematology and urinalysis. Any change in clinical laboratory abnormalities which were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: From start of study drug administration up to 24 hours post-dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

14. Secondary Outcome: Safety: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Reported as TEAEs
Description: 12-lead ECG were evaluated. Any change in ECG assessments which are deemed clinically significant by the investigator were reported as TEAEs.
Time Frame: From start of study drug administration up to 24 hours post-dose
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Participants | 0

15. Secondary Outcome: Safety: Percentage of Participants With Normal Oxygen Saturation Values Collected During Hospital Setting
Description: Oxygen saturation is the amount of oxygen that is in bloodstream and is measured as the percentage of blood hemoglobin that is carrying oxygen. Normal oxygen saturation levels are considered to be 95-100 percent; low oxygen saturation values indicate worse disease. Oxygen saturation was measured and recorded on room air. The investigator recorded the oxygen saturation as well as the oxygen delivery system and amount of oxygen administered during hospital setting. Percentage of participants with normal oxygen saturation values collected during hospital setting were reported.
Time Frame: 0.5, 1, 4, 6 and 24 hours post-dose
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | SHP615
Number analyzed (Participants) | 3
Percentage of participants | 100

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Day 8)
Arm/Group | SHP615
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP615 (N=3)
Febrile convulsion (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP615 (N=3)
Somnolence (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT03336450/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT03336450/SAP_001.pdf